CLINICAL TRIAL: NCT02832544
Title: INVestIgation of rheumatiC AF Treatment Using Vitamin K Antagonists, Rivaroxaban or Aspirin Studies
Brief Title: INVestIgation of rheumatiC AF Treatment Using Vitamin K Antagonists, Rivaroxaban or Aspirin Studies, Non-Inferiority
Acronym: INVICTUS-VKA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Population Health Research Institute (Other)
Collaborators: University of Cape Town (Other); Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: INVICTUS - VKA
Record Dates: First submitted 2015-12-10; First posted 2016-07-14 (Estimated); Last update posted 2022-10-05 (Actual); Status verified 2022-07

CONDITIONS: Rheumatic Heart Disease
Keywords: atrial fibrillation; stroke
MeSH Terms: conditions — Rheumatic Heart Disease; Atrial Fibrillation; Stroke | interventions — Rivaroxaban; acarboxyprothrombin; Warfarin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rivaroxaban (20 mg) (Experimental): Rivaroxaban 20 mg od (n ~ 2250); 15 mg od (once daily) in patients with creatinine clearance (CrCl) 15-49 ml/min
  Interventions: Drug: Rivaroxaban (20 mg)
- Vitamin K antagonists (VKA) (Active Comparator): Any approved VKA in the participating country (n ~ 2250); VKA titrated to achieve an INR of 2.0-3.0
  Interventions: Drug: Vitamin K antagonists (VKA)

INTERVENTIONS:
Drug: Rivaroxaban (20 mg) — Rivaroxaban is non-inferior to VKAs for the prevention of stroke or systemic embolism in patients with AF/flutter and RVHD and potentially superior to VKAs.
  Other Names: Xarelto
  Arms: Rivaroxaban (20 mg)
Drug: Vitamin K antagonists (VKA)
  Other Names: Warfarin
  Arms: Vitamin K antagonists (VKA)

SUMMARY:
This program is a comprehensive evaluation of rheumatic valvular heart disease (RVHD), Atrial fibrillation (AF)/flutter and stroke.

A prospective, randomized, parallel group, open-label clinical trial of rivaroxaban versus standard vitamin K antagonists (VKA) therapy to evaluate non-inferiority of rivaroxaban to VKA, with testing for superiority if non-inferiority is satisfied.

DETAILED DESCRIPTION:
Non-Inferiority Trial of rivaroxaban versus VKAs: 4,500 patients

Inclusion Criteria:

1. RVHD diagnosed by echocardiography at any time prior to enrollment
2. Age ≥18
3. Increased risk of stroke by any of the following

   1. CHA2DS2-VASc score ≥ 2 OR
   2. Moderate/Severe mitral stenosis with valve area ≤2.0 cm2 OR
   3. Left atrial spontaneous echo contrast OR
   4. Left atrial thrombus
4. Heart Rhythm a) AF or Flutter should be documented on baseline 12-lead ECG, or on a previous 12-lead ECG, Holter monitor, in-hospital ECG rhythm strip or Pacemaker or ICD electrogram.

Treatment:

Patients will be randomized either to receive rivaroxaban or any approved VKA. Treatment will be open-label.

1. Rivaroxaban Arm

   * Rivaroxaban 20 mg once daily
   * Rivaroxaban 15 mg once daily (for patients with an creatinine clearance ≥15 and <50 ml/min)
2. VKA Arm

   * Any VKA approved for use in the participating country
   * VKA titrated to achieve an INR of 2.0-3.0

ELIGIBILITY:
Inclusion Criteria:

1. RVHD diagnosed by echocardiography at any time prior to enrollment
2. Age ≥18
3. Increased risk of stroke by any of the following

   * CHA2DS2-VASc score ≥ 2 OR
   * Moderate/Severe mitral stenosis with valve area ≤2.0 cm2 OR
   * Left atrial spontaneous echo contrast OR
   * Left atrial thrombus
4. Heart Rhythm *AF or Flutter should be documented on baseline 12-lead ECG, or on a previous 12-lead ECG, Holter monitor, in-hospital ECG rhythm strip or Pacemaker or ICD electrogram.

Exclusion Criteria:

1. Refusal to give informed consent
2. Actively involved in any study that would compromise the protocol of INVICTUS Trial
3. Severe co-morbid condition with life expectancy < 1 year
4. Other serious condition(s) or logistic factors likely to interfere with study participation or with the ability to complete the trial, as appropriate to country or region.
5. Likely to have valve replacement surgery within 6 months
6. Mechanical valve prosthesis or other condition requiring treatment with VKAs. Patients with deep vein thrombosis or recent pulmonary embolism can be enrolled where both VKAs and rivaroxaban are approved.
7. Contraindication to the study medication of the trial

   * Allergy to rivaroxaban
   * Allergy to VKAs ( non-inferiority trial)
   * Allergy to aspirin ( superiority trial)
8. Severe renal insufficiency with an calculated creatinine clearance (Cockcroft-Gault) <15 ml/min
9. Serious bleeding in the past six months or at high risk for bleeding
10. Moderate to severe hepatic impairment
11. Ongoing need for dual antiplatelet therapy (patients with on-going aspirin therapy ≤100 mg per day are not excluded)
12. Ongoing need for dual strong inhibitors of CYP-3a4 or p-glycoprotein inhibitor.
13. Received an investigational drug in the past 30 days
14. Patients considered unsuitable for trial inclusion because of unwillingness to attend follow up visits
15. Women who are pregnant and/or breastfeeding
16. Women of child bearing age who do not use an effective form of birth control.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4565 (Actual)
Dates: Start 2016-08-22 (Actual); Primary Completion 2022-08-18 (Actual); Study Completion 2022-08-18 (Actual)

PRIMARY OUTCOMES:
Time from randomization to the first occurrence of vascular death or death of unknown cause, stroke, myocardial infarction or systemic embolism | Approximately 4 years
  Vascular death or death of unknown cause, stroke, myocardial infarction or systemic embolism

SECONDARY OUTCOMES:
Time from randomization to the first occurrence of composite of stroke or systemic embolism | Approximately 4 years
  Composite of stroke or systemic embolism

OTHER OUTCOMES:
Time from randomization to the first occurrence of a Major Bleed | Approximately 4 years
  using the ISTH major bleeding definition

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Connolly, MD, Principal Investigator — Population Health Research Institute
Locations (139):
- Princess Marina Hospital, Gaborone, Botswana
- Brazil (12):
  - Cardresearch - Cardiologia Assistencial e de Pesquisa, Belo Horizonte, Minas Gerais
  - Nucleo de Estudios Clinicos - Universidade Federal do Triângulo Mineiro, Uberaba, Minas Gerais
  - Eurolatino Pesquisas Médicas Ltda, Uberlândia, Minas Gerais
  - Clínica Procardio Ltda., Blumenau, Santa Catarina
  - Instituto de Pesquisa Clínica de Campinas, Campinas
  - LOEMA - Instituto de Pesquisa Clínica & Consultores Ltda, Campinas
  - Via Médica Centro Clínico Barroso e Sebba Ltda, Goiânia
  - Instituto de Cardiologia do Rio Grande do Sul, Porto Alegre
  - Fundação Faculdade de Medicina de São José do Rio Preto, São José do Rio Preto
  - Instituto do Coração - HCFMUSP, São Paulo
  - Instituto Dante Pazzanese de Cardiologia, São Paulo
  - Santa Casa de Misericórdia de Votuporanga, Votuporanga
- Cameroon (4):
  - Clinique Coeur Et Vie, Douala
  - Douala General Hospital, Douala
  - St. Elizabeth Catholic General Hospital, Cardiac Centre, Kumbo
  - Hopital Central Yaounde, Yaoundé
- China (22):
  - Liangxiang Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital/School of Clinical Medicine of Guangdong Pharmaceutical University, Guangzhou, Guangdong
  - Jixi People's Hospital, Jixi, Heilongjiang
  - Tieli People's Hospital, Yichun, Heilongjiang
  - Luoyang Central's Hospital Affiliated to Zhengzhou University, Luoyang, Henan
  - Dancheng County People's Hospital, Zhoukou, Henan
  - Suiping Renan Hospital, Zhumadian, Henan
  - Jianshi County People's Hospital, Enshi, Hubei
  - Suqian Peaple's Hospital of Nanjing Drum-Tower Hospital Group, Suqian, Jiangsu
  - Tonghua Central Hospital, Tonghua, Jilin
  - Affiliated Zhongshan Hospital of Dalian University, Dalian, Liaoning
  - The First Affiliated Hospital of Dalian Medical University, Dalian, Liaoning
  - Ningxia Peple's Hospital, Yinchuan, Ningxia
  - Pi County People's Hospital, Chengdu, Sichuan
  - Anyue County People's Hospital, Ziyang, Sichuan
  - Wendeng Central Hospital, Weihai, Wendeng
  - Ninghai People's Hospital, Ningbo, Zhejiang
  - Beijing Anzhen Hospital, Beijing
  - Zhongmou County People's Hospital, Henan
  - Zhengzhou No.7 People's Hospital, Henan
  - Zhengzhou 9th People's Hospital, Henan
  - Guangshan County People's Hospital, Henan
- Egypt (14):
  - Fayoum General Hospital, Al Fayyum
  - Mehallah Rheumatic Heart Center, Al Mansurah
  - Specialized Medical Hospital - Mansoura, Al Mansurah
  - Alexandria University Hospital, Alexandria
  - Assuit General Hospital, Asyut
  - Benha University Cardiology Department, Banhā
  - Beni Suef University Hospital, Banī Suwayf
  - Ain Shams University Hospital, Cairo
  - Kasr El Einy Hospital (Cairo University), Cairo
  - Suez Canal University Hospital, Ismailia
  - El Minia University Hospital, Minya
  - Sohag University, Sohag, Sohag
  - Red Crescent Hospital, Tanta
  - Zagazig University Hospital, Zagazig
- Ethiopia (4):
  - Hawassa University Referral Hospital, Awasa, Snnpr
  - College of Health Sciences, Addis Ababa University, Black Lion Hospital, Addis Ababa
  - Jimma University Hospital, Jimma
  - Mekelle University, Mek'ele
- India (7):
  - Sri Jayadev Institute of Cardiovascular Sciences and Research, Bangalore, Karnataka
  - Dr. Ram Manohar Lohia Hospital @ PGIMER, New Delhi, National Capital Territory of Delhi
  - Govind Ballabh Pant Hospital (GIPMER), New Delhi, National Capital Territory of Delhi
  - All India Institute of Medical Sciences, New Delhi, National Capital Territory of Delhi
  - SMS Medical College, Jaipur, Rajasthan
  - King George's Medical College, Lucknow, Uttar Pradesh
  - Sanjay Gandhi Post Graduate Institute of Medical Sciences, Lucknow, Uttar Pradesh
- Kazakh National Medical Institute,, Almaty, Kazakhstan
- Kenya (3):
  - Moi Teaching and Referral Hospital, Eldoret
  - Karen Hospital, Nairobi
  - Kenyatta National Hospital / University Of Nairobi, Nairobi
- Clinical Hospital of administrative department of President and Government of Kyrgyz Republic, Bishkek, Kyrgyzstan
- Malawi (3):
  - Queen Elizabeth Central Hospital, Blantyre
  - Kumuzu Central Hospital, Lilongwe
  - Mzuzu Central Hospital, Mzuzu
- Mexico (7):
  - Hospital Angeles León, León, Guanajuato
  - Hospital Bernardette, Guadalajara, Jalisco
  - Centro de Estudios Clínicos de Querétaro S.C., Querétaro City, Querétaro
  - Centro para el Desarrollo de la Medicina y Asistencia Especializada S.C., Culiacán, Sinaloa
  - Instituto de Investigación del Hospital Cardiológica Aguascalientes, Aguascalientes
  - Hospital General Dr. Jorge Soberon Acevedo.Secretaria de Salud del Estado de Guerrero, Guerrero
  - Instituto Nacional de Cardiología Ignacio Chavez, México
- Mozambique (2):
  - Maputo Central Hospital, Maputo
  - Instituto Nacional de Saude & Universidade Eduardo Mondlane, Maputo
- Nepal (9):
  - College of Medical Sciences, Bharatpur
  - Chitwan Medical College, Bharatpur
  - Nobel medical college and teaching hospital pvt ltd, Biratnagar
  - Gautam Buddha Community Heart Hospital, Butwāl
  - BP Koirala Institute of Health Sciences, Dharān
  - Manmohan Cardiothoracic Vascular and Trasplant Center, IOM, TU, Kathmandu
  - Sahid Gangalal Heart Center, Kathmandu
  - Bheri Zonal Hospital, Nepalgunj
  - Manipal College of Medical Sciences, Pokhara
- Nigeria (9):
  - Federal Medical Center, Abeokuta
  - University of Nigeria Teaching Hospital, Enugu
  - College of Medicine, University of Ibadan, Ibadan
  - Jos University Teaching Hospital, Jos
  - Ahmadu Bello University Teaching Hospital, Kaduna
  - Aminu Kano University Teaching Hospital, Kano
  - Department of Medicine, Lagos University Teaching Hospital, Lagos
  - Ladoke Akintola University of Technology Teaching Hospital, Ogbomoso
  - Department of Medicine, Delta State University Teaching Hospital, Oghara
- Pakistan (5):
  - Punjab Institute of Cardiology, Lahore, Punjab Province
  - Isra University Hospital, Hyderābād
  - Nishtar Hospital Multan, Multan
  - Lady Reading Hospital, Peshawar
  - Rawalpindi Institute of Cardiology, Rawalpindi
- Paraguay (5):
  - Instituto Nacional de Cardiología, Asunción
  - Hospital Barrio Obrero, Asunción
  - Hospital Regional de Ciudad Del Este, Ciudad del Este
  - Hospital Nacional Itaugua, Itauguá
  - Clinical Hospital, San Lorenzo
- Philippines (4):
  - Palawan Medical City, Puerto Princesa City, Palawan
  - Philippine General Hospital, Manila
  - Philippine Heart Center, Quezon City
  - Quirino Memorial Medical Center, Quezon City
- University of Rwanda, Kigali University Teaching Hospital, Kigali, Rwanda
- South Africa (8):
  - Nelson Mandela Academic Hospital, Mthatha, Eastern Cape
  - Charlotte Maxeke Academic Hospital, Johannesburg, Parktown
  - Sefako Makgatho Health Sciences University, Ga-Rankuwa, Pretoria
  - Cardiology Research Universitas private hospital, Bloemfontein
  - University of Cape Town, Cape Town
  - University of Limpopo, Polokwane
  - Port Elizabeth Hospital Complex, Port Elizabeth
  - Chris Hani Baragwanath Hospital, Soweto
- Sudan (8):
  - Alobeid Teaching Hospital, Al-Ubayyid
  - Atbara Teaching Hospital, Atbara
  - Ahmed Gasim Hospital, Khartoum
  - Alshaab Teaching Hospital, Khartoum
  - Ahmed Gasim Pediatric Hospital, Khartoum
  - Sudan Heart Center, Khartoum
  - Digna Prince Hospital, Port Sudan
  - Medani Heart Centre, Wad Medani
- Tanzania (2):
  - Muhimbili University of Health and Allied Sciences, Dar es Salaam
  - Mbeya Zonal Referral Hospital, Mbeya
- Uganda Heart Institute, Kampala, Uganda
- Zambia (3):
  - Livingstone Central Hospital, Livingstone
  - University Teaching Hospital (UTH), Lusaka
  - Ndola Central Hospital, Ndola
- Zimbabwe (3):
  - Mpilo Hospital, National University Science & Technology, Bulawayo
  - Harare Hospital, Harare
  - Parirenyatwa Hospital, Harare

IPD SHARING:
Plan to Share IPD: No
cumulative participant data only

REFERENCES:
- [Derived] Connolly SJ, Karthikeyan G, Ntsekhe M, Haileamlak A, El Sayed A, El Ghamrawy A, Damasceno A, Avezum A, Dans AML, Gitura B, Hu D, Kamanzi ER, Maklady F, Fana G, Gonzalez-Hermosillo JA, Musuku J, Kazmi K, Zuhlke L, Gondwe L, Ma C, Paniagua M, Ogah OS, Molefe-Baikai OJ, Lwabi P, Chillo P, Sharma SK, Cabral TTJ, Tarhuni WM, Benz A, van Eikels M, Krol A, Pattath D, Balasubramanian K, Rangarajan S, Ramasundarahettige C, Mayosi B, Yusuf S; INVICTUS Investigators. Rivaroxaban in Rheumatic Heart Disease-Associated Atrial Fibrillation. N Engl J Med. 2022 Sep 15;387(11):978-988. doi: 10.1056/NEJMoa2209051. Epub 2022 Aug 28. PMID 36036525
- [Derived] Karthikeyan G, Connolly SJ, Yusuf S. Overestimation of Stroke Risk in Rheumatic Mitral Stenosis and the Implications for Oral Anticoagulation. Circulation. 2020 Nov 3;142(18):1697-1699. doi: 10.1161/CIRCULATIONAHA.120.050347. Epub 2020 Nov 2. No abstract available. PMID 33136507
- [Derived] Karthikeyan G, Connolly SJ, Ntsekhe M, Benz A, Rangarajan S, Lewis G, Yun Y, Sharma SK, Maklady F, Elghamrawy AE, Kazmi K, Cabral TTJ, Dayi H, Changsheng M, Gitura BM, Avezum A, Zuhlke L, Lwabi P, Haileamlak A, Ogah O, Chillo P, Paniagua M, ElSayed A, Dans A, Gondwe-Chunda L, Molefe-Baikai OJ, Gonzalez-Hermosillo JA, Hakim J, Damasceno A, Kamanzi ER, Musuku J, Davletov K, Connolly K, Mayosi BM, Yusuf S; INVICTUS Investigators. The INVICTUS rheumatic heart disease research program: Rationale, design and baseline characteristics of a randomized trial of rivaroxaban compared to vitamin K antagonists in rheumatic valvular disease and atrial fibrillation. Am Heart J. 2020 Jul;225:69-77. doi: 10.1016/j.ahj.2020.03.018. Epub 2020 Mar 25. PMID 32474206